CLINICAL TRIAL: NCT00080210
Title: A Phase II Study of Multiple Doses of Intravenous Puricase in Subjects With Hyperuricemia and Refractory Gout
Brief Title: A Study of Persons With Gout Who Do Not Respond to or Are Allergic to Conventional Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Savient Pharmaceuticals (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C0403
Record Dates: First submitted 2004-03-24; First posted 2004-03-25 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Gout
Keywords: elevated uric acid; Elevated serum uric acid level; Symptomatic gout
MeSH Terms: conditions — Gout | interventions — Pegloticase

INTERVENTIONS:
Drug: Puricase

SUMMARY:
This is a randomized, open-label, multicenter, parallel-groups study of multiple intravenous doses of Puricase, administered intravenously, in 40 patients with symptomatic gout. Subjects must wash out of any uric acid-lowering agents for one week before being dosed, and must refrain from using such agents throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Subjects to be included in the study are:

* Outpatients of either gender, age 18 or older
* Diagnosed with symptomatic gout refractory to conventional therapy or unable to tolerate conventional therapy (for example: having one or more tophi and/or having experienced a gout flare within the previous 6 months and/or having chronic, gouty arthritis)
* Hyperuricemic: screening serum uric acid must be >=8 mg/dL.
* The patient must be willing and able to give informed consent and adhere to visit/protocol schedules (Consent must be given before any study procedures are performed)
* Women of childbearing potential must have a negative serum pregnancy test and must use an approved birth control method during their participation in the protocol. Such methods include oral, injectable, or implantable contraceptives; IUDs and barrier contraceptives in combination with spermicide

Exclusion Criteria:

Subjects to be excluded are those for whom any of the following apply:

* Unstable coronary artery disease or uncontrolled hypertension
* History of end stage renal disease requiring dialysis
* History of liver disease, as defined by baseline serum transaminase elevation >3X the upper limit of normal in the absence of any other known cause
* Organ transplant recipient requiring immunosuppressive therapy
* Concurrent use of prednisone at a dose >10 mg qd (or equivalent) at or within one week before dosing
* Concurrent use of uric acid-lowering agents
* Prior treatment with Puricase® or other recombinant uricase
* An acute gout flare within one week prior to first treatment with Puricase® (exclusive of chronic synovitis/arthritis) requiring use of medication which violates the protocol
* glucose-6-phosphate dehydrogenase deficiency
* A history of anaphylactic reaction to a recombinant protein or porcine derivatives
* Lactation
* Has taken an investigational drug within 4 weeks prior to study drug administration or plans to take an investigational agent during the study
* Known allergy to urate oxidase or PEGylated products
* Has any other medical or psychological condition which, in the opinion of the investigator, might create undue risk to the patient or interfere with the patient's ability to comply with the protocol requirements

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-03; Study Completion 2005-02

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Spain Rehabilitation Center, Birmingham, Alabama
  - University of California, San Diego, La Jolla, California
  - University of Chicago Dept of Medicine, Chicago, Illinois
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - Center for Rheumatology and Bone Research, Wheaton, Maryland
  - North Shore University Hospital Division of Rheumatology, Manhasset, New York
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health & Science University Arthritis & Rheumatic Diseases, Portland, Oregon
  - Pride Clinical research Associates, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Sundy JS, Becker MA, Baraf HS, Barkhuizen A, Moreland LW, Huang W, Waltrip RW 2nd, Maroli AN, Horowitz Z; Pegloticase Phase 2 Study Investigators. Reduction of plasma urate levels following treatment with multiple doses of pegloticase (polyethylene glycol-conjugated uricase) in patients with treatment-failure gout: results of a phase II randomized study. Arthritis Rheum. 2008 Sep;58(9):2882-91. doi: 10.1002/art.23810. PMID 18759308